CLINICAL TRIAL: NCT01972256
Title: Prospective Multicenter Clinical Evaluation of Fusion
Brief Title: A Study Comparing Fusion Rates of Two Lumbar Fusion Procedures
Status: Completed | Type: Observational
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-0023
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Pseudoarthrosis; Spinal Stenosis; Spondylolisthesis; Degenerative Disc Disease (DDD)
MeSH Terms: conditions — Pseudarthrosis; Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Previous transsacral fusion: Subject candidates are those who had required a transsacral fusion at L4-L5-S1 where these were the only lumbar levels treated for pseudoarthrosis, spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD).
- Previous transforaminal lumbar interbody fusion: Subject candidates are those who had required transforaminal lumbar interbody fusion at L4-L5-S1 where these were the only lumbar levels treated for pseudoarthrosis, spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD).

SUMMARY:
The purpose of this study is to demonstrate the relative efficacy of two lumbar fusion procedures: transacral lumbar interbody fusion when used in conjunction with unilateral or bilateral posterior pedicle screw fixation as an adjunct to fusion, in comparison to transforaminal lumbar interbody fusion (TLIF) when used in conjunction with unilateral or bilateral supplemental screw fixation as an adjunct to fusion.

Subject candidates are those who had previously required and received fusion at L4-L5-S1 where these were the only lumbar levels treated for pseudoarthrosis, spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD).

DETAILED DESCRIPTION:
Consecutive subjects who were treated with the transsacral lumbar interbody fusion or TLIF procedures at least 2 years prior to the date the data is collected will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Male or female subject that had previously received the transsacral two-level procedure when used in conjunction with pedicle screw or facet screw fixation or TLIF two-level procedure with unilateral or bilateral supplemental screw fixation (e.g. pedicle screws, facet screws at L4-L5-S1 to treat pseudoarthrosis, spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD)
* Subject that was treated no less than 2 years prior to this evaluation with an transsacral or TLIF procedure by the participating surgeons
* Subject that had a diagnosis that required a transsacral or TLIF procedure at the L4-L5-S1 levels and did not require treatment at any other lumbar levels at the time of surgery

Exclusion Criteria:

* Subject who did not receive the transsacral or TLIF procedure for fusion of L4-L5-S1
* Subject who received lumbar fusion procedures at levels other than L4-L5-S1 at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject candidates are those who had required fusion at L4-L5-S1 where these were the only lumbar levels treated for pseudoarthrosis, spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Efficacy | Assessed at 2 years post-op or greater
  Fusion of the targeted vertebral bodies (L4-L5-S1) at 24 months as determined by independent orthopedic surgeon reviewer interpretation of high resolution Computed Tomography (CT) scan.

SECONDARY OUTCOMES:
Safety | 2 years post-op
  Incidence of major device-related adverse events and/or failures, defined as those requiring revision surgery or a secondary operation, or events resulting in permanent disability or death.

OTHER OUTCOMES:
Additional Secondary Endpoint: Efficacy | Assessed at 2 years post-op
  Comparative Lordosis of L4-S1 at 24-months as determined by an independent orthopedic surgeon reviewer's interpretation of 24-month lateral (neutral) radiographs compared to baseline.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Indiana Spine Group, Indianapolis, Indiana
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Michigan Spine Institute, Waterford, Michigan
  - Brazos Spine, College Station, Texas